CLINICAL TRIAL: NCT05792007
Title: Etude du Microenvironnement médullaire Dans Les Leucémies Aiguës de l'Enfant
Brief Title: Study of the Medullary Microenvironment in Acute Childhood Leukemia
Acronym: MILA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: DR220254-MILA; 2022-A02570-43 (Registry Identifier: IdRCB)
Record Dates: First submitted 2023-03-08; First posted 2023-03-30 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Acute Lymphoid Leukemia; Acute Myeloid Leukemia in Children
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Intervention Model Description: Open-label, interventional monocentric biological study in two parallel and controlled groups
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with acute leukemias (Active Comparator): Children with acute lymphoid leukemia B, acute lymphoid leukemia -T or acute myeloid leukemia
  Interventions: Procedure: Biological sampling in patients
- Control group (Other): Children without blood diseases
  Interventions: Procedure: Biological sampling in control patients

INTERVENTIONS:
Procedure: Biological sampling in patients — blood and bone marrow samples from patients with Acute Leulemia.
  Arms: Patients with acute leukemias
Procedure: Biological sampling in control patients — blood and bone marrow samples from children undergoing orthopedic surgery exposing the bone marrow.(osteotomy of the pelvis).
  Arms: Control group

SUMMARY:
Acute leukemia (AL) is the most common cancer in children. Despite the optimization of chemotherapy treatments and the development of supportive care, a certain number of LAs relapse and/or progress to death of the child. It therefore seems essential to try to better understand the physiopathology and the mechanisms of resistance to treatment of these diseases.

DETAILED DESCRIPTION:
Acute leukemia (AL) is the most common cancer in children. Despite the optimization of chemotherapy treatments and the development of supportive care, a certain number of AL's relapse and/or progress to death of the child. It therefore seems essential to try to better understand the physiopathology and the mechanisms of resistance to treatment of these diseases. The study of the microenvironment appears in this context as a promising avenue. The bone marrow microenvironment is composed of an extracellular matrix and cells, in particular mesenchymal stromal stem cells (MSC's). In adult acute leukemia, it has been clearly demonstrated that these microenvironment cells are reprogrammed by leukemia cells to allow the development and proliferation of the latter. Links have also been demonstrated in acute leukemia between the cells of the microenvironment and resistance to chemotherapy. In a certain number of cases, the support of the microenvironment for the development of leukemia or resistance to chemotherapy involves modulation of the energy metabolism of leukemia cells. This notably involves interactions between leukemic cells and MSCs and re-programming of the energy metabolism of the latter. To date, there are only very few studies concerning the role of the microenvironment in acute childhood leukemia and none to date has specifically studied the energy metabolism (oxidative phosphorylation and glycolysis) of MSCs.

ELIGIBILITY:
Inclusion Criteria:

* for patients with AL:

  1. Child with acute lymphoblastic or myeloblastic leukemia at diagnosis
  2. Not having received prior hematological treatment
  3. Aged 1 to 15 years old
  4. Whose 2 parents, or the holder of parental authority, have signed a consent enlightened.
  5. Affiliated patient or beneficiary of a social security scheme.
* Control group patients:

  1. Child undergoing orthopedic surgery exposing the bone marrow (osteotomy of the pelvis).
  2. Aged between 1 and 15 years old.
  3. Having no pathology of hematological origin.
  4. Not having received any treatment that could interfere with the functioning of the bone marrow.
  5. Whose 2 parents or the holder of parental authority have signed a consent enlightened.
  6. Affiliated patient or beneficiary of a social security scheme.

Exclusion Criteria:

* for patients with AL:

  1. Patient under 1 year old and over 15 years old.
  2. Contraindication to myelogram.
  3. Absence of signature of the informed consent by the 2 parents or the holder of parental authority.
  4. Patients with relapsed acute lymphoblastic or myeloblastic leukemia.
  5. Having received prior hematological treatments.
  6. Parents with physical or mental condition not allowing to understand the informed consent.
* Control group patients

  1. Patient under 1 year old and over 15 years old.
  2. Having an underlying haematological pathology.
  3. Absence of signature of the informed consent by the 2 parents or the holder of parental authority.
  4. Having received prior hematological treatments.
  5. Parents with physical or mental condition not allowing to understand informed consent.

Ages: 1 Year to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2023-10-26 (Actual); Primary Completion 2026-10-25 (Estimated); Study Completion 2028-10-24 (Estimated)

PRIMARY OUTCOMES:
Oxygen Consumption Rate | At inclusion
  Difference in oxidative phosphorylation measured by OCR (Oxygen Consumption Rate) in pmol/min/nd DNA between the mesenchymal stromal stem cells (MSCs) of children with Acute Leukemia and those of children without blood diseases.

SECONDARY OUTCOMES:
Difference in Extra Cellular Acidification Rate | At inclusion
  Difference in glycolysis, measured by the ECAR (Extra Cellular Acification Rate) in mpH/min/ng DNA between the MSCs of children with AL and those of children without hematological disease.
Difference in Reactive Oxygen Species | At inclusion
  Difference in oxidative metabolism thanks to the measurement of reactive oxygen species (ROS), measured in MIF/isotype, between MSCs of children with AL and those of children without hematological disease
Difference in doubling time in culture | At inclusion
  The difference in doubling time in culture (measured in days) between the MSCs of children with LA and those of children free of hemopathy. At each passage, the number of living and dead MSCs will be counted.
Difference in Immunophenotypic profile | At inclusion
  The difference in immunophenotypic profile (cytometry, immunofluorescence) between MSCs of children with AL and those of children without hematological disease. Use of a panel of monoclonal antibodies directed against various membrane antigens (CD45, CD34, CD14, CD90, CD73, CD105).
Difference in mutational profiles between MSCs and leukemia cells | At inclusion
  Difference in mutational profiles between MSCs and leukemia cells from children with AL. Comparison of mutations acquired by leukemic cells compared to stromal cells by an NGS-type high-throughput sequencing approach.
Differences in transcriptomic signatures between MSCs and MSC subpopulations | At inclusion
  Differences in transcriptomic signatures between MSCs and MSC subpopulations of children with AL and those of children without hematological disease. The RNAs of the MSCs obtained after culture will be extracted then reverse-transcribed into cDNA. The quality control of the extracted RNAs will be carried out on a Bioanalyzer (Agilent). Transcriptome analysis of the MSC pool will be performed by RNA Seq/NGS. Transcriptomic identification of MSC subpopulations will be performed by single-cell RNAseq/NGS.
Differences in cytokine profiles within the bone marrow | At inclusion
  Differences in cytokine profiles in the bone marrow and in the blood, measured in ng/mL, between children with AL and children without hematological disease.ELISA-like assay of IL-3, IL-6, IL-7, IL-8, IL-10, IL-15, TGF-bêta, IFN-gamma

CONTACTS AND LOCATIONS:
Overall Officials: Olivier HERAULT, MD-PhD, Study Director — University Hospital of TOURS; Julien LEJEUNE, MD-PhD, Principal Investigator — University Hospital of TOURS
Locations (3):
- France (3):
  - Service d'hématologie biologique-CHRU TOURS, Tours
  - Service d'onco-hématologie pédiatrique -CHRU Tours, Tours
  - Service de chirurgie orthopédique pédiatrique -CHRU TOURS, Tours

IPD SHARING:
Plan to Share IPD: No